CLINICAL TRIAL: NCT03122522
Title: A Phase II Study to Evaluate Adaptive Dosing of Ipilimumab and Nivolumab Combination Immunotherapy
Brief Title: A Study to Evaluate Adaptive Dosing of Ipilimumab and Nivolumab Combination Immunotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-162
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Melanoma
Keywords: unresectable; III or stage IV; Ipilimumab; Nivolumab; 17-162
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ipilimumab and nivolumab (Experimental): Pts will receive 2 doses of ipilimumab 3mg/kg + nivolumab 1mg/kg every 3 weeks. Week 6, if pts have achieved a favorable antitumor effect by RECIST will begin maintenance nivolumab alone at 480mg every 4 weeks for 2 doses (week 6 & week 10) & repeat response assessments at week 12. If pts don't achieve a favorable antitumor effect at week 6, pt will get 2 additional doses of ipilimumab + nivolumab every 3 weeks & then will be assessed for response at week 12. If pts haven't achieved a favorable antitumor effect by week 12, if felt in the best interest for the pt as determined by the PI, pts may continue getting additional doses of ipilimumab + nivolumab with response reassessments after every 2 doses. Maintenance nivolumab will continued until unacceptable toxicity or confirmed disease progression. If pts have had an initial clinical benefit from therapy & subsequently experience progressive disease at any time, reinduction with combination ipilimuma+ nivolumab will be allowed.
  Interventions: Drug: ipilimumab; Drug: nivolumab

INTERVENTIONS:
Drug: ipilimumab — ipilimumab 3mg/kg
Drug: nivolumab — nivolumab 1mg/kg

SUMMARY:
This study will help determine whether 2 doses of the combination (ipilimumab + nivolumab) is sufficient for patients with early benefit compared to the usual way of trying to give 4 doses. If patients do not show early benefit after 2 doses, patients will be able to continue with additional ipilimumab + nivolumab, even beyond the standard 4 doses if felt in the best interest of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of unresectable III or stage IV metastatic melanoma.
* Subjects must have at least 1 extracranial, unresectable, non-bony lesion that is measurable radiographically (based on RECIST 1.1).
* No prior CTLA-4 or PD-1/PD-L1 therapy for the treatment of metastatic disease.
* ECOG performance status of 0-1.
* Life expectancy ≥ 4 months.
* Screening laboratory parameters:

  * White blood cell (WBC) count ≥ 2000/μL;
  * Absolute neutrophil count (ANC) ≥ 1500/μL;
  * Platelets ≥ 100,000/μL;
  * Hemoglobin (Hgb) ≥ 9 g/dL;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN);
  * Total bilirubin ≤ 1.5 × ULN (< 3 mg/dL for subjects with Gilbert's disease);
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below): Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL] Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL]
* Age ≥ 18 years.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for 23 weeks after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

[Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).] Nonsterilized males who are sexually active with a female partner of childbearing potential must use 2 acceptable methods of effective contraception from Day 1 and for 31 weeks after receipt of the final dose of investigational product.

Acceptable methods of effective contraception are described in the following table:

* Barrier Methods - Male condom plus spermicide, cap plus spermicide, or diaphragm plus spermicide.
* Intrauterine Device Methods-Copper T, or Levonorgestrel-releasing intrauterine system (e.g., Mirena®), also considered a hormonal method.
* Hormonal Methods-Implants, hormone shot or injection, combined pill, minipilimumabll, or Patch.

Exclusion Criteria:

* Active autoimmune disease or any condition requiring systemic treatment with either corticosteroids (>10 mg daily of prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* History of motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre Syndrome, Myasthenia Gravis).
* Other active, concurrent malignancy that requires ongoing systemic treatment or interferes with radiographic assessment of melanoma response as determined by the investigator.
* Known immunodeficiency or HIV, Hepatitis B, or Hepatitis C infection. Antibody to Hepatitis B or C without evidence of active infection may be allowed.
* History of severe allergic reactions to any unknown allergens or any components of the study drugs.
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for immunological and clinical assessments or post-study follow-up contact to determine relapse and survival.
* Women who are breastfeeding or who are pregnant as evidenced by a positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) performed within 14 days of the first dose of study drug and by a urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours of the first dose of study drug(s).
* Any condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
objective response rate | at 6 weeks
  RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Postow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (14):
  - Hartford Healthcare Alliance (Data Collection Only), Hartford, Connecticut
  - Jaykumar Thumar, Hartford, Connecticut
  - JOHNS HOPKINS HOSPITAL (Data Analysis Only), Baltimore, Maryland
  - Brigham and Women's Hospital (Data and Specimen Analysis Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Hospital for Special Surgery (Data Analysis), New York, New York
  - Columbia University (Data Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pandit-Taskar N, Mauguen A, Frosina D, Jungbluth A, Busam KJ, Lyashchenko S, Schwartz J, Momtaz P, Warner AB, Smithy JW, Shoushtari AN, Callahan MK, Chapman PB, Postow MA. Programmed death ligand-1 PET imaging in patients with melanoma: a pilot study. Melanoma Res. 2025 Oct 1;35(5):328-338. doi: 10.1097/CMR.0000000000001050. Epub 2025 Jun 25. PMID 40557547
- [Derived] Postow MA, Goldman DA, Shoushtari AN, Betof Warner A, Callahan MK, Momtaz P, Smithy JW, Naito E, Cugliari MK, Raber V, Eton O, Nair SG, Panageas KS, Wolchok JD, Chapman PB. Adaptive Dosing of Nivolumab + Ipilimumab Immunotherapy Based Upon Early, Interim Radiographic Assessment in Advanced Melanoma (The ADAPT-IT Study). J Clin Oncol. 2022 Apr 1;40(10):1059-1067. doi: 10.1200/JCO.21.01570. Epub 2021 Dec 20. PMID 34928709
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm